CLINICAL TRIAL: NCT05452551
Title: Investigation of Myotonometer Reliability in Evaluation of Plantar Fascia Biomechanical Properties in Individuals With Diabetes
Brief Title: Investigation of Myotonometer Reliability in Evaluation of Plantar Fascia Biomechanical Properties
Status: Completed | Type: Observational
Sponsor: İlke KARA, PT (Other)
Collaborators: Bitlis Eren University (Other); Medipol University (Other)
Responsible Party: Sponsor-Investigator, İlke KARA, PT, Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: BEU-IK-02
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Diabetes Mellitus; Plantar Fascia
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Myotonometric measurement — MyotonPRO is a non-invasive myotonometer used to evaluate the viscoelastic properties of soft tissues. Data collection will be carried out by three researchers experienced in the use of myotonometer. Before the evaluations, participant and repeated measurement information for both researchers will be recorded on the device. All assessments will be made bilaterally. The first researcher will perform two measurements 30 minutes apart from the measurement point standardized with MyotonPRO to evaluate the plantar mechanical properties. Then, the second researcher will take two measurements with MyotonPRO from the same point with 30 minutes intervals. One day later, the first researcher will measure again from the same reference point once.

SUMMARY:
The study aims to examine the intra-rater, inter-rater, and inter-session reliability of MyotonPRO in measuring plantar fascia mechanical properties in adults with diabetes.

DETAILED DESCRIPTION:
Therefore, changes occur in standing weight-bearing points, loading zones, and gait biomechanics. The thickened plantar fascia increases the risk of developing diabetic foot with increased peak-plantar pressure, and therefore, plantar fasciitis is more common in individuals with diabetes than in healthy individuals. The myotonometer studies showed that chronic diabetes history increases dynamic stiffness, which is one of the mechanical properties of the plantar fascia, and that as the severity of the disease increases, fascial stiffness also increases. The aim of the study is to examine the intra-rater, inter-rater, and inter-session reliability of MyotonPRO in measuring plantar fascia mechanical properties in adults with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body mass index < 30 kilogram/meter square
* Willing to participate in the study
* Diagnosed with Type 2 Diabetes
* HbA1c level ≥ 6.5% mmol/mol
* Fasting plasma glucose ≥126 mg/dl
* Random plasma glucose ≥ 200 mg/d

Exclusion Criteria:

* History of lower extremity injuries
* Ulceration localized on plantar fascia
* Age ≥ 65 years
* Any use of medication that will affect muscle tone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between 18-35 years old diagnosed with Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Muscle Tone (Hz) | Day 1
  The muscle tone which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. After each application, the acceleration graph will be examined and if there is any deviation from the normal, the measurements will be repeated. Recordings will be reloaded into the software program and reported for each participant. The oscillation frequency (Hz) represents the resting muscle tone.
Stiffness (N/m) | Day 1
  The muscle tone which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. After each application, the acceleration graph will be examined and if there is any deviation from the normal, the measurements will be repeated. Recordings will be reloaded into the software program and reported for each participant.
Logarithmic decrement | Day 1
  The muscle tone which is a biomechanical property of the forearm muscles will be evaluated with a portable hand-held myotonometer. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph. After each application, the acceleration graph will be examined and if there is any deviation from the normal, the measurements will be repeated. Recordings will be reloaded into the software program and reported for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Çevik Saldıran, PhD, Study Director — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No